CLINICAL TRIAL: NCT06588101
Title: Clinical Trial Recruitment and Retention Strategies for Family Members in the Intensive Care Unit: A Study Within A Trial Randomized Design
Brief Title: Clinical Trial Recruitment and Retention Strategies for Family Members in the ICU
Acronym: SWAT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: 2024-4023
Record Dates: First submitted 2024-04-19; First posted 2024-09-19 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Family Members; Recruitment; Clinical Study; Retention; Recruitment of Participants; Study Enrollment; Retention of Participants; Compensation Incentives
MeSH Terms: interventions — Compensation and Redress

STUDY DESIGN:
Intervention Model Description: 2x2 Design for randomization strategies 2x2 Desgin for retention strategies
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Both recruitment strategies (Experimental): Consent form with Infographic + Large compensation
  Interventions: Other: Written informed consent with infographic; Other: Compensation
- Neither recruitment strategy (No Intervention): Consent form + No compensation
- One recruitment strategy - Infographic (Experimental): Consent form with Infographic + No compensation
  Interventions: Other: Written informed consent with infographic
- One recruitment strategy - Compensation (Experimental): Consent form + Large compensation
  Interventions: Other: Compensation

INTERVENTIONS:
Other: Written informed consent with infographic — Potential participants are provided a visual infographic depicting the key elements of the written consent form in addition to the standard written consent form.
  Arms: Both recruitment strategies; One recruitment strategy - Infographic
Other: Compensation — Potential participants are provided an e-gift card to Amazon or Second Cup as a reward for completing the enrollment questionnaire.
  Arms: Both recruitment strategies; One recruitment strategy - Compensation

SUMMARY:
There is a need to identify strategies that improve the conduct of clinical trials involving family members of intensive care unit (ICU) patients. The purpose of the present study is to evaluate recruitment and retention strategies for clinical trials involving family members of ICU patients. 4 strategies (2 recruitment and 2 retention) will be tested. Investigators will integrate the strategies into three existing studies that involve family members of ICU patients. Participants will be randomized using a 2x2 factorial design. The co-primary outcomes are recruitment percentage (participants enrolled/participants approached) and retention percentage (participants completing follow-up/participants enrolled).

DETAILED DESCRIPTION:
Family engagement in the ICU is recommended by critical care professional societies, but insufficient evidence of its benefits for patients and family members has hindered clinical uptake. Thus, high-quality evidence is needed to promote and support family engagement practices. A specific unmet need is to identify strategies to improve the recruitment and retention of families in clinical trials in the ICU setting. The objective of this study is to evaluate recruitment and retention strategies for clinical trials involving family members in the ICU setting.

Methodological Approach: Investigators will use a Study Within a Trial (SWAT) design to embed a factorial randomized trial of 160 participants enrolled across investigator group's three ongoing studies involving family members of ICU patients: FAME, VR-Family, and NGAGE. Investigators expect 160 participants to be enrolled over a 6-month period. Participants will be randomized by 2x2 factorial design to selected recruitment and/or retention strategies. The co-primary outcomes will be (1) recruitment rate and (2) retention rate.

ELIGIBILITY:
Inclusion Criteria:

* Has family member admitted to an intensive care unit.
* Expected hospital stay > 48 hours
* Able to participate in English or French

Exclusion Criteria:

* Has another family member participating in the trial
* Repeat admissions within the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment percentage | At enrolment
  Family member participants enrolled/ family member participants approached
Retention percentage | From enrolment until 6 month follow-up completion
  Family member participant completing follow-up/family member participants enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD, MSc, Principal Investigator — Lady Davis Institute, McGill University, Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No